CLINICAL TRIAL: NCT06206850
Title: Neo-Bio-ADAURA: a Single Arm, Multi-Centre Phase II Study to Evaluate Mechanisms of Resistance to Neoadjuvant Osimertinib.
Brief Title: Neo-Bio-ADAURA: a Phase II Study to Evaluate Mechanisms of Resistance to Neoadjuvant Osimertinib
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jair Bar, M.D., Ph.D. (Other Government)
Responsible Party: Sponsor-Investigator, Jair Bar, M.D., Ph.D., Deputy Director - Institute of Oncology. Head of Thoracic Oncology Unit, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-21-21629
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-01

CONDITIONS: Non-squamous NSCLC
Keywords: NSCLC; Resectable; EGFR; stage II-III
MeSH Terms: interventions — osimertinib

STUDY DESIGN:
Intervention Model Description: Single arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant osimertinib (Experimental): Osimertinib 80 mg QD
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Oral Osimertinib 80 mg once daily (QD) for the duration of 9 weeks (3 cycles).
  Other Names: Tagrisso

SUMMARY:
This study is a single-arm phase II study of neoadjuvant osimertinib as monotherapy for the treatment of patients with resectable stage II-III non-small cell lung cancer (NSCLC) harboring an epidermal growth factor receptor (EGFR) sensitizing mutation (L858R or deletion in exon 19 [Ex19del]).

DETAILED DESCRIPTION:
This study is a single-arm phase II study of neoadjuvant osimertinib as monotherapy (or in combination with chemotherapy-to be considered only if the interim analysis of the ongoing NeoADAURA study would indicate futility of single-agent osimertinib) for the treatment of patients with resectable stage II-III non-small cell lung cancer (NSCLC) harboring an epidermal growth factor receptor (EGFR) sensitizing mutation (L858R or deletion in exon 19 [Ex19del]). Twenty subjects will be included in the study. Potential participants diagnosed with resectable (clinical stage II to IIIB) NSCLC will undergo pre-screening to identify if they carry an EGFR common mutation (Ex19del and/or L858R) - histologically or cytologically. Eligible subjects will receive neoadjuvant osimertinib 80 mg monotherapy once daily (QD) for 9 weeks (3 cycles) followed by surgery (Note: neoadjuvant osimertinib in combination with chemotherapy- will be considered only if the interim analysis of the ongoing NeoADAURA study would indicate futility of single-agent osimertinib). Osimertinib will be continued up to surgery. After surgery, outside of the study protocol the subjects may continue receiving osimertinib 80 mg QD for three years as adjuvant therapy (per local reimbursement), and/or other adjuvant therapy according to relevant standard of care (SoC; platinum + pemetrexed) until disease progression or death. The subjects will be followed up for safety (30 days after the surgery as part of the current protocol's assessments) and survival status (data to be collected as part of SOC, up to 5 years after the last dose of osimertinib).

Tumour specimens will be used for correlative studies to identify molecular mechanisms of tumour resistance to treatment. If available, formalin-fixed paraffin embedded (FFPE) tumour biopsies will be collected at baseline. Resected tumour specimens will be collected during surgery. When possible, recurrence FFPE tumour biopsies will also be collected.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent for the trial prior to any study specific procedures. The subject must also provide consent for correlative translational study.
* Male or female subjects who are ≥18 years of age on the day of signing the informed consent.
* Histologically or cytologically documented non-squamous NSCLC with completely resectable (Stage II-III) disease.

Note: thick needle biopsy of endobronchial ultrasound (EBUS)/bronchoscopy is acceptable.

* Complete surgical resection of the primary NSCLC must be deemed achievable, as assessed by a multi-disciplinary team evaluation (which should include a thoracic surgeon, specialised in oncologic procedures).
* Performance status (ECOG) 0-1 at enrolment, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing.
* Lung function test results allowing curative surgery by thoracic surgeon's assessment.
* Cardiac function by ECHO cardiography results allowing curative surgery by thoracic surgeon's assessment.
* Have adequate normal organ and marrow function, including the following:

  * Absolute neutrophil count ≥1.5×109/L.
  * Platelet count ≥ 100×109/L.
  * Haemoglobin ≥ 9.0 g/dL. Note: The use of granulocyte colony stimulating factor (G-CSF) support, platelet transfusion and blood transfusions to meet these criteria is not permitted.
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 times the upper limit of normal (ULN).
  * Total bilirubin (TBL) ≤1.5 times the ULN or for patients with documented/suspected Gilbert's disease, bilirubin ≤2 times the ULN.
  * Creatinine ≤1.5 times the ULN or creatinine clearance ≥50 mL/min (creatinine clearance can be measured or calculated by Cockcroft and Gault equation). If neoadjuvant chemotherapy is part of the neoadjuvant treatment regimen3, calculated creatinine clearance must be ≥60 mL/min.
* Body weight >30 kg.
* Life expectancy of >6 months prior to enrolment.
* A tumour which harbours one of the 2 common EGFR mutations known to be associated with EGFR-TKI sensitivity (Ex19del, L858R), either alone or in combination with other EGFR mutations (ie, T790M, G719X, S7681 and L861Q). Exon 20 insertion co-mutation are not permitted.
* Female patients who are not abstinent (in line with the preferred and usual lifestyle choice of the patient) and intend to be sexually active with a male partner must use highly effective contraceptive measures. Women of child-bearing potential must have a negative urine or serum pregnancy test within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required prior to the first dose of any study treatment if they are of child-bearing potential; or must have evidence of non-child-bearing potential by fulfilling 1 of the following criteria at screening:

  * Post-menopausal, defined as 50 years of age or more and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
  * Women under 50 years old would be considered as postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and have luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the post-menopausal range for the institution.
  * Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation (Further information is available in Appendix B (Definition of Women of Childbearing Potential and Acceptable Contraceptive Methods).
* Male patients must be willing to use barrier contraception.

Exclusion Criteria:

* Known active infection with hepatitis C virus (HVC) or tuberculosis. Patients positive for HCV antibody are eligible only if the polymerase chain reaction is negative for HCV RNA. Screening for chronic conditions is not required.
* Known active or uncontrolled infection with hepatitis B virus (HBV) (i.e., known positive HBV surface antigen [HBsAg] result).

Participants with HBV infection may be included only if they meet all the following criteria:

* Demonstrated absence of HCV co-infection or history of HCV co-infection
* Demonstrated absence of HIV infection
* Participants with active HBV infection are eligible if they are:

  * Receiving anti-viral treatment for at least 6 weeks prior to study treatment
  * HBV DNA is suppressed to <100 IU/mL
  * transaminase levels are below ULN.
* Participants with a resolved or chronic infection HBV are eligible if they are:

  * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc IgG].
  * Receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment and 6-12 months (to be determined by a hepatologist) post-treatment or
  * Positive for HBsAg, but for >6 months have had transaminases levels below ULN and HBV DNA levels below <100 IU/mL (i.e., are in an inactive carrier state).
  * Receiving anti-viral prophylaxis for 2-4 weeks prior to study treatment and 6-12 months (to be determined by a hepatologist) post-treatment.

    * HIV active infection (e.g. patients receiving treatment for infection)

Should participants with HIV infection be included, patients are only eligible if they meet all the following criteria:

* Undetectable viral RNA load for 6 months
* CD4+ count of >350 cells/μL
* No history of AIDS-defining opportunistic infection within the past 12 months'
* Stable for at least 4 weeks on the same anti-HIV medications

  * Past medical history of interstitial lung disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically significant ILD.
  * A history of another primary malignancy, except for the following:

    * Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of osimertinib and of low potential risk for recurrence
    * Adequately treated non-melanoma skin cancer or lentigo malignancy without evidence of disease
    * Adequately treated carcinoma in situ without evidence of disease.
  * Has pre-operative radiotherapy treatment as part of the care plan.
  * Refractory nausea and vomiting, chronic gastrointestinal diseases causing inability to swallow osimertinib, or previous significant bowel resection that would preclude adequate absorption of osimertinib.
  * Mixed small cell and NSCLC histology.
  * T4 tumours infiltrating the aorta, the oesophagus and/or the heart; and/or any bulky N2 disease.
  * Any of the following cardiac criteria:

    * Mean resting corrected QT interval (QTc) > 470 msec obtained from 3 electrocardiograms (ECGs), using the screening clinic ECG machine-derived QTcF value
    * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECG, e.g., complete left bundle branch block, second-degree heart block, and third-degree heart block.
    * Patient with any factors that increase the risk of QTc prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including serum/plasma potassium below the lower limit of normal [LLN]; serum/plasma magnesium <LLN; serum/plasma calcium <LLN , congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes (TdP).
  * Currently pregnant (confirmed with positive pregnancy test) or breast-feeding.
  * Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment with the exception of alopecia and grade 2 prior platinum-therapy related neuropathy.
  * Prior treatment (within the previous 12 months) with any systemic anti-cancer therapy for NSCLC including chemotherapy, biologic therapy, immunotherapy, hormonal therapy or any investigational drug/product.
  * Prior treatment (within the previous 12 months) with EGFR-TKI therapy.
  * Current use of medications or herbal supplements known to be strong inducers of cytochrome P450(CYP)3A4, or unable to stop use of such medications at least 3 weeks prior to receiving the first dose of study treatment.
  * Ongoing treatment with immune suppressing drugs (e.g., methotrexate for rheumatoid disease, continuous systemic steroids for chronic obstructive pulmonary disease, etc.).
  * Any major surgical procedure (as defined by the Investigator) which occurred within 28 days prior to the first dose of osimertinib. Procedures such as placement of vascular access, biopsy via mediastinoscopy or biopsy via video-assisted thoracoscopic surgery (VATS) are permitted.
  * Involvement in the planning or conduct of the study (applies to both Investigator staff and/or staff at the study site).
  * Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater.
  * Concurrent enrolment in another clinical study, unless it is an observational (noninterventional) clinical study or during the follow-up period of an interventional study.
  * Prior randomization or treatment in a previous osimertinib clinical study regardless of treatment arm assignment.
  * Previous enrolment in the present study.
  * Known allergy or hypersensitivity to any of the study drugs, study drug excipients, drugs with a similar chemical structure or class, or anaesthetics.
  * Inability of the patient, in the opinion of the investigator, to understand and/or comply with study medications, procedures and/or follow-up OR any conditions that, in the opinion of the investigator, may render the patient unable to complete the study.
  * Any condition that, in the opinion of the Investigator, would interfere with the evaluation of patient safety or study results, including, but not limited to, ongoing or active infection, uncontrolled hypertension, active bleeding diatheses, unstable angina pectoris, significant cardiac arrhythmia, interstitial lung disease, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs from study treatment, or compromise the ability of the patient to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Identification of mechanisms of resistance to EGFR in surgical specimens | Up to approximately 5 years
  Identification of mechanisms of resistance to osimertinib (alone or in combination with chemotherapy), based on assessment of the post-osimertinib surgical specimens.
Frequency of various resistance mechanisms to EGFR | Up to approximately 5 years
  The proportion of cells harbouring each mechanism within each tumour.
Identify mechanisms of resistance to EGFR in surgical specimens | Up to approximately 5 years
  Mechanisms that correlate with different levels of pathologic response.

SECONDARY OUTCOMES:
Evaluate the efficacy of neoadjuvant osimertinib for resectable EGFR mutant NSCLC per rate of pathological complete response (pCR) | Up to approximately 5 years
  Absence of all cancer cells in the tumor after completion of neoadjuvant treatment with Osimertinib.
Evaluate the efficacy of neoadjuvant osimertinib for resectable EGFR mutant NSCLC per major pathologic response (MPR) | Up to approximately 5 years
  10% or less viable tumour cells.
Rate of pathological downstaging | Up to approximately 5 years
  Downstaging will be is assessed in accordance with the AJCC 8th edition TNM staging system. Pathological downstaging is defined as baseline N2 patients becoming N1/N0 or N1 to N0 at the time of surgery, and/or downstaging of T-stage at surgery.
Event-free survival (EFS defined as time to disease progression that precludes surgery, disease recurrence or death of any cause) of treated patients. | Up to approximately 5 years
  Defined as time to disease progression that precludes surgery, disease recurrence or death of any cause of treated patients. 1, 3 and 5-year EFS rate of treated patients.
Overall survival (OS) of treated patients | Up to approximately 5 years
  1, 3 and 5-year OS rate of treated patients.
Rate of R0 resection | Up to approximately 5 years
  Rate of R0 resection will be described by percentages with 95% CI (by Wilson).

CONTACTS AND LOCATIONS:
Locations (2):
- Israel (2):
  - Sheba Medical Center, Ramat Gan, Israel
  - Sheba Medical Center, Jusidman Cancer Center, Ramat Gan, Israel

IPD SHARING:
Plan to Share IPD: No